CLINICAL TRIAL: NCT07194252
Title: The Effect of Guided Imagery Applied Before and After Surgery on Surgical Anxiety, Pain, and Analgesic Consumption in Patients Undergoing Total Joint Arthroplasty: A Randomized Controlled Trial
Brief Title: The Effect of Guided Imagery Technique on Anxiety, Pain, and Analgesic Use in Total Joint Arthroplasty Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, BTuran, Lecturer, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: YBU-HEM-RK-01
Record Dates: First submitted 2025-09-10; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Total Joint Arthroplasty
Keywords: pain; anxiety; analgesic; total joint arthroplasty
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention Grubs (Experimental): The intervention group's surgical anxiety levels were assessed using the "Surgical Anxiety Scale" during the preoperative period. Subsequently, at the relevant clinic, the scale was administered twice on the day before the scheduled surgery date (at noon and in the evening) and once each at 48 and 72 hours post-surgery, for a total of four times. At the end of the application, the "Surgical Anxiety Scale" and the "Surgical-Specific Anxiety Scale" will be reapplied to the intervention group. In the postoperative period, participants' pain intensity will be measured using the "NRS" at 48 hours postoperatively before the intervention, immediately after the intervention, and at 72 hours before the intervention and immediately after the intervention.
  Interventions: Other: Guided imagery technique application
- Control Grubs (No Intervention): During the preoperative period, nursing care will be provided according to the routine care protocol of the clinic where the study is conducted. Subsequently, participants' levels of surgical anxiety will be assessed using the "Anxiety Scale Specific to Surgery" simultaneously with the intervention group patients. In the postoperative period, participants' pain intensity will be measured using the "NRS" at 48 and 72 hours postoperatively and will be measured again 60 minutes after the measurements (simultaneously with the intervention group patients). In the final stage, the analgesic consumption of the intervention and control groups will be evaluated on the 2nd and 3rd days of the postoperative period using the "Analgesic Consumption Tracking Form" to assess the administration status of the analgesic drugs included in the treatment protocol, and the application phase of the study will be completed.

INTERVENTIONS:
Other: Guided imagery technique application — Intervention is a guided imagery technique designed for patients undergoing total joint arthroplasty. It will be administered in a total of 4 sessions: once daily on the day before surgery, twice daily on the day of surgery, and once daily on the 2nd and 3rd days after surgery, accompanied by imagery scenarios developed in accordance with the Compact Disc (CD) and literature developed by the Turkish Psychological Association. The study aims to examine its effects on surgical anxiety levels, postoperative pain intensity, and analgesic consumption. This approach is structured as a non-pharmacological method specific to surgical nursing practice and differs from previous similar studies in that it is applied in both the preoperative and postoperative periods using the same sample in the literature.
  Arms: intervention Grubs

SUMMARY:
This randomized controlled study will investigate the effects of guided imagery on preoperative anxiety and postoperative pain and analgesic consumption in patients undergoing total joint arthroplasty. Conducted between September 2025 and June 2026 at a public hospital in Zonguldak, Turkey, the study will include patients scheduled for total joint arthroplasty following ethics committee approval. The intervention group will receive guided imagery twice preoperatively and once daily at 48 and 72 hours postoperatively. Outcomes will be assessed using the Surgical Anxiety Scale, surgery-specific anxiety scale, Numerical Rating Scale (NRS), and analgesic consumption tracking.

DETAILED DESCRIPTION:
This study aimed to investigate the effects of preoperative guided imagery on anxiety and postoperative guided imagery on pain intensity and analgesic consumption in patients undergoing total joint arthroplasty. This randomized controlled trial (RCT) study's population consisted of patients undergoing total joint arthroplasty at the Orthopedics and Traumatology Clinic of a public hospital in Zonguldak province between September 2025 and June 2026. The required sample size and power calculations for this study were performed using the G*Power program, with an effect size of 0.76 for the independent samples t-test. The minimum number of participants to provide 80% test power at a 95% confidence level was 58 for each surgical group, totaling 116 participants. The following data collection tools will be used: a "Descriptive Patient Information Form," a "Surgical Anxiety Scale," a "Surgery-Specific Anxiety Scale," a "Numerical Rating Scale (NRS)," and an "Analgesic Consumption Tracking Form." In the first stage, the "Descriptive Patient Information Form" will be administered to both the intervention and control groups. Then, surgical anxiety levels will be assessed using the "Surgical Anxiety Scale" and the "Surgery-Specific Anxiety Scale" in both the intervention and control groups. Guided imagery will then be administered to the intervention group twice preoperatively (in the afternoon and evening) one day before the scheduled surgery date and once at the 48th and 72nd hours postoperatively. At the end of the intervention, the "Surgical Anxiety Scale" and the "Surgery-Specific Anxiety Scale" will be administered again to the intervention group. In the postoperative period, the pain intensity of the intervention group will be measured with the "NRS" at the 48th and 72nd postoperative hours, before and immediately after the intervention. The surgical anxiety levels of the control group patients will be assessed simultaneously with the intervention group using the "Surgical Anxiety Scale" and "Surgery-Specific Anxiety Scale" without any intervention. In the postoperative period, the pain intensity of the control group will be measured with the "NRS" at the 48th and 72nd postoperative hours and will be measured again after these measurements simultaneously with the intervention group. Finally, the analgesic consumption of the intervention and control groups will be assessed on the 2nd and 3rd postoperative days using the "Analgesic Consumption Tracking Form," concluding the intervention phase. Microsoft-Excel 2019 and International Business Machines (IBM) Statistical Package for the Social Sciences (SPSS) 22.0 will be used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone unilateral arthroplasty surgery,
* Without cognitive impairment,
* Who speak and write Turkish,
* Without hearing or vision problems,
* Without any other acute illness causing pain or anxiety,
* Who received the same analgesic agent in the treatment protocol during the postoperative period,
* And who volunteered to participate in the study will be included.

Exclusion Criteria:

* Having a diagnosis of chronic pain syndrome or neuropathic pain,
* Having a diagnosis of psychiatric illness/being under treatment
* Continuous use of analgesic/sedative medication that may affect the pain threshold,
* Hearing impairment or severe cognitive impairment that prevents participation in guided imagery applications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2026-05-22 (Estimated); Study Completion 2026-06-22 (Estimated)

PRIMARY OUTCOMES:
Surgical Anxiety Scale | September 2025-June 2026 (9 months)
  The scale was developed in Turkish by Karanci and Dirik (2003) and is a 5-point Likert-type scale (1: Strongly disagree, 5: Strongly agree). The scale consists of 10 statements covering fears that patients may experience regarding surgery. The maximum score that can be obtained from the scale is 50. High scores on the scale reflect anxiety about experiencing pain, dying during surgery, and complications and restrictions that may arise after surgery. The Cronbach's Alpha coefficient for the scale was found to be 0.79.

SECONDARY OUTCOMES:
Numerical Rating Scale | September 2025-June 2026 (9 months)
  The NRS is a single-dimensional scale that uses 11 numbers (ranging from 0 to 10) to measure pain intensity. The patient is asked to select the number that best reflects their pain intensity, where 0 = no pain and 10 = the worst (unbearable) pain. The NRS has been shown to be a valid and reliable measurement tool for assessing postoperative acute pain intensity in adults and the elderly, as well as in elderly patients with mild to moderate cognitive impairment, and is widely used in clinical and research settings.
Analgesic Consumption Tracking Form | September 2025-June 2026 (9 months)
  This form is used to evaluate analgesic consumption on the 2nd and 3rd days after surgery for patients in the intervention and control groups to examine the effect of guided imagery on analgesic consumption in the postoperative period. This form, created by the researcher, aims to inquire about and compare the analgesic agent used, the dose, the method and frequency of administration, and the analgesic agent used in case of need in the intervention and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay YAZICI, Assoc. Prof., Study Director — Ankara Yildirim Beyazıt University
Locations (1):
- Zonguldak Atatürk State Hospital, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT07194252/Prot_SAP_000.pdf
  • Informed Consent Form (2025-09-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT07194252/ICF_001.pdf